CLINICAL TRIAL: NCT05700422
Title: A Single-arm Investigator Initiated Study to Evaluate the Efficacy of OC-01 (Varenicline Solution) Nasal Spray on Signs and Symptoms of Dry Eye Disease in Subjects With Sjogren's Syndrome
Brief Title: Nasal Spray Study in Sjogren's Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Principal Investigator, Giacomina Massaro-Giordano, Clinician, Co-Director, Penn Dry Eye & Ocular Surface Center, and Professor of Clinical Ophthalmology, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 851655
Record Dates: First submitted 2023-01-14; First posted 2023-01-26 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Sjogren's Syndrome; Dry Eye
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- OC-01 (varenicline solution) 0.03 mg nasal spray (Experimental)
  Interventions: Drug: Varenicline Nasal Spray

INTERVENTIONS:
Drug: Varenicline Nasal Spray — OC-01 (varenicline solution) 0.03 mg nasal spray

SUMMARY:
This study will investigate how well OC-01 (varenicline) nasal spray can treat the signs and symptoms of dry eye disease in those Sjogren's Syndrome. Patients at least 18 years old with moderate-to-severe Sjogren's dry eye disease may be eligible for this study. If you are eligible to participate in the study and you decide to join, there will be 3 study visits over approximately 1 month. You will also self-administer the nasal spray at home every day, 2 times a day during this month.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written consent prior to study-related procedures
* Be at least 18 years of age at the screening visit
* Have diagnosed moderate to severe Sjogrens Syndrome via blood work or biopsy Category 2 staining score for Conjunctiva based on the Van Bjisterveld and Utrect scale and 3 staining score for cornea based on the NEI scale
* Have been using Cyclosporine or Lifitegrast 3 months
* Be literate and able to complete questionnaires independently
* Be able and willing to use the study drug and participate in all study assessments and visits
* Have sufficient hand strength, in the opinion of the Investigator, to be able to independently administer the study drug
* Have provided verbal and written informed consent
* If a female is of childbearing potential, they must: use an acceptable means of birth control (acceptable methods of contraception include: hormonal oral, implantable, injectable, or transdermal contraceptives, mechanical spermicide in conjunction with a barrier such as a diaphragm or condom, IUD, or surgical sterilization of partner), and have a negative urine pregnancy test on Day 1

Exclusion Criteria:

Have undergone previous ocular surgery (e.g., intraocular, oculoplastic, corneal or refractive surgical procedure)

* Have had thermal pulsation or IPL in prior 3 months
* Have used topical ophthalmic corticosteroid therapy in prior 4 weeks
* Have had cataract surgery in the last 6 months
* Have clinically significant ocular trauma.
* Have active ocular Herpes simplex or Herpes Zoster infection
* Have ocular inflammation (uveitis, iritis, scleritis, episcleritis, keratitis, conjunctivitis) at the discretion of the investigator.
* Have ocular infection (e.g., viral, bacterial, mycobacterial, protozoan or fungal infection or the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids including hordeolum/stye).
* Have retinal pathology that can limit visual potential and refractive outcomes in the opinion of the investigator
* Have severe (Grade 3 or 4) inflammation of the eyelid (e.g., blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis)
* Have eyelid abnormalities that significantly affect the lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis).
* Have ocular surface abnormality that may compromise the corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, map dot fingerprint dystrophy, or the effect of any other ophthalmic medication that might in the opinion of the investigator compromise the ocular surface integrity).
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Have chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the Investigator, may lead to clinically significant risk of increased bleeding.
* Have had nasal or sinus surgery (including history of application of nasal cautery) or significant trauma to these areas
* Be currently treated with nasal continuous positive airway pressure
* Have any untreated nasal infection at Visit 1
* Have a vascularized polyp, severely deviated septum, chronic recurrent nosebleeds, or severe nasal obstruction as confirmed by intranasal examination performed at Visit 1.
* Have a known hypersensitivity to any of the procedural agents or study drug components
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to Visit 1 and during the treatment period.
* Be a female who is pregnant, nursing, or planning a pregnancy at Visit 1. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal oral, implantable, injectable, or transdermal contraceptives; mechanical spermicide in conjunction with a barrier such as a diaphragm or condom; IUD; or surgical sterilization of partner. The risks of OC-01 among pregnant patients are not known.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Scheie Eye Institute at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gupta AS, Linaburg TJ, Iacobucci E, Augello PA, Qin VL, Ying GS, Bunya VY, Massaro M. Varenicline Solution Nasal Spray for the Treatment of Dry Eye Disease in Sjogren's Disease: A Pilot Study. Clin Ophthalmol. 2025 Mar 27;19:1073-1084. doi: 10.2147/OPTH.S512364. eCollection 2025. PMID 40166690

RESULTS

PARTICIPANT FLOW:
Groups:
- OC-01 (Varenicline Solution) 0.03 mg Nasal Spray: Varenicline Nasal Spray: OC-01 (varenicline solution) 0.03 mg nasal spray every 12 hours
Period: Overall Study
Arm/Group | OC-01 (Varenicline Solution) 0.03 mg Nasal Spray
Started | 39
Completed | 35
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | OC-01 (Varenicline Solution) 0.03 mg Nasal Spray
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Cornea Staining
Description: The National Eye Institute (NEI) scale is the method that will be used to measure corneal staining using fluorescein strips on a scale of 0-3. The scale is a density-based scoring from 0-3 with 0 indicating no staining and 3 indicating highest density of staining.
Time Frame: Baseline to Day 28
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OC-01 (Varenicline Solution) 0.03 mg Nasal Spray
Number analyzed (Participants) | 35
units on a scale | -1.78 [-2.09 to -1.47]

2. Primary Outcome: Mean Change in Eye Dryness Score as Measured by the Visual Analogue Scale (VAS)
Description: VAS is a validated, subjective measure for acute and chronic pain. Patients rate eye dryness on a scale of 0-100 where 0 corresponds to "no discomfort" and 100 corresponds to "maximal discomfort."
Time Frame: Baseline to Day 28
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OC-01 (Varenicline Solution) 0.03 mg Nasal Spray
Number analyzed (Participants) | 35
score on a scale | -14.51 [-25.60 to -3.41]

3. Primary Outcome: Mean Change in Conjunctival Staining
Description: The Van Bijsterveld and Utrecht scale is the method that will be used to measure conjunctival staining while using lissamine green dye. The scale is a from 0-3 with 0 indicating no staining and 3 indicating confluent staining.
Time Frame: Baseline to Day 28
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OC-01 (Varenicline Solution) 0.03 mg Nasal Spray
Number analyzed (Participants) | 35
units on a scale | -0.46 [-0.91 to -0.01]

4. Secondary Outcome: Mean Change in Best Corrected Visual Acuity
Description: LogMAR or Logarithm of the Minimum Angle of Resolution was the method used for measuring best correct visual acuity (BCVA). LogMAR is a scale from -0.2 to 1.6 where the letter size is described in LogMAR units such that LogMAR -0.2 is equivalent to 20/12 (best vision) and LogMAR 1.6 is equivalent to 20/800 (Worse vision). The letter size change in units of 0.1 LogMAR from one row to the next.
Time Frame: Baseline to Day 28
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | OC-01 (Varenicline Solution) 0.03 mg Nasal Spray
Number analyzed (Participants) | 35
logMAR | 0.01 [-0.04 to 0.05]

5. Secondary Outcome: Mean Change in Dry Mouth Scale
Description: VAS is a validated, subjective measure for acute and chronic pain. Patients rate mouth dryness on a scale of 0-100 where 0 corresponds to "no discomfort" and 100 corresponds to "maximal discomfort."
Time Frame: Baseline to Day 28
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OC-01 (Varenicline Solution) 0.03 mg Nasal Spray
Number analyzed (Participants) | 35
units on a scale | -9.58 [-20.52 to 1.35]

6. Secondary Outcome: Mean Change in Nose Dryness Scale
Description: VAS is a validated, subjective measure for acute and chronic pain. Patients rate nose dryness on a scale of 0-100 where 0 corresponds to "no discomfort" and 100 corresponds to "maximal discomfort."
Time Frame: Baseline to Day 28
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | OC-01 (Varenicline Solution) 0.03 mg Nasal Spray
Number analyzed (Participants) | 35
units on a scale | -0.44 [-11.16 to 12.05]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over the 1 month of each participants enrollment.
Arm/Group | OC-01 (Varenicline Solution) 0.03 mg Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 22/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OC-01 (Varenicline Solution) 0.03 mg Nasal Spray (N=39)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT05700422/Prot_SAP_000.pdf